CLINICAL TRIAL: NCT07064993
Title: Intraoperative and Postoperative Effects of Tramadol and Dexamethasone Added to Washing Solution in Knee Arthroscopies
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Arzu Esen Tekeli, Associate Professor Doctor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 19.11.2024
Record Dates: First submitted 2025-02-10; First posted 2025-07-15 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Nausea and Vomitting; VAS Will be Used to Assess Pain Postoperative; Itching; Chills
Keywords: Knee arthroscopy; analgesia; general anesthesia
MeSH Terms: conditions — Nausea; Pruritus; Chills; Agnosia | interventions — Observation

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, controlled, double-blind,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Standart knee arthroscopy washing solution was used. No drugs administered
  Interventions: Other: Observation
- study group (Experimental): 100 mg tramadol + 8 mg dexamethasone will be added to each 1000cc washing solution of the patients in the study group. (tramadol max i.v dose: 400 mg/day) dexamethasone max i.v dose: 32 mg/day)
  Interventions: Procedure: Experimental

INTERVENTIONS:
Other: Observation — Routine monitoring and observation
  Arms: Control group
Procedure: Experimental — Administration of tramadol and dexmethasone to arthroscopy solution
  Arms: study group

SUMMARY:
To evaluate the effects of tramadol and dexamethasone added to washing solutions on postoperative nausea and vomiting, VAS score, itching and chills in knee arthroscopy cases.

Randomised, double-blind, prospective, clinical trial

Research Question(s):

1. Do tramadol and dexamethasone added to the washing solution have any effect on postoperative parameters in knee arthroscopy cases?
2. Does the postoperative efficacy change depending on the dose of tramadol and dexamethasone in the washing solution?

Translated with DeepL.com (free version)

DETAILED DESCRIPTION:
Knee arthroscopy is a minimal surgical treatment method that allows closed intervention under anaesthesia for the diagnosis and treatment of joint disorders. The natural structure of the joints is preserved as much as possible and no unnecessary tissue damage is caused. The most important advantage is the possibility to reach every part of the joint and provide complete treatment.The aim of the study was to evaluate the effects of tramadol and dexamethasone added to washing solutions on postoperative nausea and vomiting, VAS score, itching and chills in knee arthroscopy cases.

Patients who are decided to undergo knee arthroscopy will be evaluated preoperatively by the anaesthesia outpatient clinic. Necessary information will be given and consent will be obtained. Patients will be randomised into 2 groups as study (S) and control (C) groups.

Study Group (Group S): 100 mg tramadol + 8 mg dexamethasone will be added to each 1000cc washing solution.

(tramadol max iv dose: 400 mg/day) (Dexamethasone max iv dose: 32mg/day) No any drugs will be used for control group solution For postoperative analgesia, 15mg/kg paracetamol iv will be administered to both groups as standard before extubation. The moment of being admitted to the PACU and having a RAMSAY sedation scale of 3 or less will be accepted as hour 0; 0, 3 and 6 hours VAS, nausea, vomiting, itching and chills will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All elective arthroscopy cases performed under general anaesthesia
* ASA 1-2 status
* Patients giving written consent

Exclusion Criteria:

* ASA 3 and above status
* Pregnant
* Cases with advanced hepatic and renal insufficiency
* Cases with bleeding diathesis
* Cases with BMI>35
* Cases requiring regional anaesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-08-02 (Estimated); Study Completion 2026-09-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain measurement | 3 hours interval
  Visual Analogue Scale scores (0 to 10, 0:no pain, 10 worst)

SECONDARY OUTCOMES:
ıntraoperative and post operative effects except VAS scores | 3 hours interval
  Non invasive blood pressure (mmHg),

CONTACTS AND LOCATIONS:
Overall Officials: Şükran Sevimli, PhD, Study Chair — Van Yuzuncu Yil University Ethics
Locations (1):
- Van Yuzuncu Yil University School of Medicine Department of Anesthesiology and Reanimation, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Personal data of the participants will be protected